CLINICAL TRIAL: NCT03611465
Title: Creation of a Pace-mapping Atlas on Healthy and Pathological Hearts
Acronym: ATLAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Dr Jean-Marc SELLAL, Cardiologist specialised in rhythmology, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-A01857-46
Record Dates: First submitted 2018-03-26; First posted 2018-08-02 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Ventricular Tachycardia
Keywords: Sudden cardiac death; Electrophysiologic exploration; Myocardial infarction
MeSH Terms: conditions — Tachycardia, Ventricular; Death, Sudden, Cardiac; Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: There is no randomization. Patients are provided into 3 groups according to their pathology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VT ablation group (Other): patients presenting history of myocardial infarction and ventricular tachycardia undergoing a VT ablation
  Interventions: Other: Standard pace-mapping examination
- pre implantation group (Experimental): patients presenting history of myocardial infarction but without history of ventricular tachycardia. Patients scheduled for a cardiac defibrillator implantation in primary prevention.
  Interventions: Other: Pace-mapping
- control group (Experimental): patients without history of myocardial infarction and without history of ventricular tachycardia, undergoing an ablation in the left atrium for an atrial fibrillation or an accessory pathway ablation.
  Interventions: Other: Pace-mapping

INTERVENTIONS:
Other: Pace-mapping — Acquire pace-mapping on three distinct populations to better understand the influence of heart disease on electrical conduction.
  Arms: control group; pre implantation group
Other: Standard pace-mapping examination — Acquire pace-mapping on three distinct populations to better understand the influence of heart disease on electrical conduction.
  Arms: VT ablation group

SUMMARY:
Aim of this study is to collect data from pace mapping performed in three groups of patients : patients presenting ventricular tachycardia and infarction history, patients presenting infarction history without presenting ventricular tachycardia, and in patients without structural heart disease.

DETAILED DESCRIPTION:
Ventricular tachycardia (VT) represent an important problem in western countries. 350 000 deaths are attributable to ventricular arrhythmias in Europe every year. The gold standard treatment is to implant a cardiac defibrillator that will be able to stop arrhythmia by delivering pacing or internal shocks.

In order to avoid internal shocks, ablation techniques have been developed, consisting in placing catheters in the left ventricle, to induce the VT, and then to perform a mapping of its circuit. Once this circuit is clearly defined, ablation of the critical part of the circuit, so called VT isthmus can be performed, using a radiofrequency power. One of the limitations of this technique is that it requires VT induction during the procedure, and that the VT lasts long enough to enable its mapping.

Nancy University Hospital developed a technique using pace mapping to define the VT isthmus even when the VT is not sustained. The pace mapping technique enables to reveal conduction troubles in the studied ventricles, that correspond with the VT isthmus.

During this study, the investigators will collect pace-mapping data from ventricles of patient presenting infarction history and VT, from patients with infarction history without VT, and from patients without ventricular pathology.

ELIGIBILITY:
Inclusion Criteria:

* Presenting one of these conditions :
* patients undergoing a VT ablation and myocardial infarction history
* patients with myocardial infarction history without VT history
* patients without myocardial infarction history but undergoing an invasive procedure in left atrium (atrial fibrillation or accessory pathway ablation)

Exclusion Criteria:

* pregnancy
* LVEF (left ventricular ejection fraction ) <20 %
* hemorrhagic stroke history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2018-10-26 (Actual); Primary Completion 2023-10-26 (Estimated); Study Completion 2024-04-26 (Estimated)

PRIMARY OUTCOMES:
Complete electrophysiology datasets for each group | the electrophysiological exploration is carried out the day after the patient's hospitalization and the datasets are generated just after removing the catheter from the patient, ie about 3 hours later the beginning of the exploration
  Collection of all complete electrophysiology datasets for each group. A data set consists of the electro-anatomical data generated by the Carto system and ECG data collected during topo-stimulation.
  Collection of all complete electrophysiology datasets for each group. A data set consists of the electro-anatomical data generated by the Carto system and ECG data collected during pace-mapping.
  It will be considered complete if 100 measurement points have been acquired (pace-mapping and ECG), covering all 17 segments of the left ventricle.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Nancy, France

REFERENCES:
- [Background] de Chillou C, Groben L, Magnin-Poull I, Andronache M, MagdiAbbas M, Zhang N, Abdelaal A, Ammar S, Sellal JM, Schwartz J, Brembilla-Perrot B, Aliot E, Marchlinski FE. Localizing the critical isthmus of postinfarct ventricular tachycardia: the value of pace-mapping during sinus rhythm. Heart Rhythm. 2014 Feb;11(2):175-81. doi: 10.1016/j.hrthm.2013.10.042. PMID 24513915